CLINICAL TRIAL: NCT02424656
Title: Alterations in the Brain's Connectome in Severe Traumatic Brain Injury
Brief Title: Alterations in the Brain's Connectome After Severe Traumatic Brain Injury
Acronym: ABCinTBI
Status: Completed | Type: Observational
Sponsor: Danish Research Centre for Magnetic Resonance (Other)
Collaborators: University of Milan (Other); University of Kiel (Other); Glostrup University Hospital, Copenhagen (Other); Lundbeck Foundation (Other); Danish Council for Independent Research (Other); Region Capital Denmark (Other)
Responsible Party: Principal Investigator, Hartwig R. Siebner, Professor, Head of research, Danish Research Centre for Magnetic Resonance
Other Study IDs: H-4-2013-186
Record Dates: First submitted 2015-04-16; First posted 2015-04-23 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Traumatic Brain Injury; Disorders of Consciousness
MeSH Terms: conditions — Brain Injuries, Traumatic; Consciousness Disorders | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Patients with TBI and DOC.
  Experimental measures (MRI, TMS-EEG, and clinical scales) will be performed at 4 time points: within 2 weeks of admission, 6-10 weeks after admission, at discharge, 1-year follow-up after TBI episode. FDG-PET will be performed in a subset of 25 patients at 3 time points: at admission, at discharge, and at 1-year follow-up.
  Interventions: Procedure: MRI; Procedure: TMS-EEG; Procedure: FDG-PET; Other: Clinical scales
- 2: Healthy patient-matched controls.
  Experimental measures (MRI, TMS-EEG, and FDG-PET) will be performed at 2 time points: within patient admission, and within patient discharge.
  Interventions: Procedure: MRI; Procedure: TMS-EEG; Procedure: FDG-PET

INTERVENTIONS:
Procedure: MRI — EEG-functional MRI, structural MRI, diffusion MRI
  Other Names: Magnetic Resonance Imaging
Procedure: TMS-EEG — Single pulse TMS combined with EEG, resting-state EEG, noise masking (auditory stimulation), electrical stimulation
  Other Names: Transcranial Magnetic Stimulation-Electroencephalogram
Procedure: FDG-PET
  Other Names: [18F]-fluorodeoxyglucose positron emission tomography
Other: Clinical scales — Evaluation of DOC: Coma recovery scale-Revised (CRS-R) and Rancho Los Amigos Scale (RLAS). Evaluation of function: Functional Independent Measure (FIMTM), and Early Functional Assessment (EFA).
  Groups: 1

SUMMARY:
This study explores the changes in whole-brain connectivity that occur during recovery from severe Traumatic Brain Injury and how these changes are related to the recovery of consciousness. Multimodal neuroimaging techniques will be used in a longitudinal fashion while patients are undergoing neurorehabilitation and after one-year of the TBI episode.

DETAILED DESCRIPTION:
Severe Traumatic Brain Injury (TBI) can result in a long-lasting altered state of consciousness. At present, the underlying neurological determinants of recovery in patients with disorders of consciousness (DOC) after a severe TBI are not well understood, and individual prognosis is very limited. Moreover, the rate of misdiagnosis between different states of altered consciousness by standard clinical scales is high, which further impacts on the clinical prognosis. In this project, multimodal neuroimaging measures will be applied and whole-brain data will be obtained from patients recovering from severe TBI in a longitudinal fashion. Patients will be examined at four time points during the sub-acute stage: immediately after admission to the neurorehabilitation unit, after ten weeks of admission, at discharge, and after one year of the TBI episode. Brain connectivity will be assessed with functional Magnetic Resonance Imaging (fMRI) combined with electroencephalography (EEG), structural MRI, diffusion MRI, high-density EEG (hdEEG) alone, and hdEEG combined with Transcranial Magnetic Stimulation (EEG-TMS), and [18F]-fluorodeoxyglucose positron emission tomography (FDG-PET).

The overall aim of the study is to find reliable biomarkers for the recovery of consciousness based on changes in cortico-cortical and cortico-subcortical brain connectivity. In order to explore this, patients that suffered a severe TBI as well a matched healthy participants group will be included in the study.

ELIGIBILITY:
Patient's inclusion criteria:

- closed-head injury

Patient's exclusion criteria:

* high level of consciousness after coma
* ventricular shunt for hydrocephalus
* large intracerebral hemorrhages or infarctions
* structural lesions in the brain stem
* locked-in syndrome due to motor pathway lesions
* contraindications for MR
* contraindications for TMS

Healthy participant's inclusion criteria:

- no prior history of neurological disorders and / or head injury

Healthy participant's exclusion criteria:

* contraindications for MR
* contraindications for TMS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. 30 Patients that have suffered a close-head TBI with associated DOC and that are admitted to neurorehabilitation at the TBI unit of Glostrup Hospital.
  2. 20 Healthy participants without history of neurological disorders, age-, gender-, and socioeconomically-matched to the included patients.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2014-09; Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Changes in whole brain connectivity as a measure of recovery of consciousness | up to 32 months

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Research Centre for Magnetic Resonance, Copenhagen, Denmark

REFERENCES:
- [Background] Conde V, Andreasen SH, Petersen TH, Larsen KB, Madsen K, Andersen KW, Akopian I, Madsen KH, Hansen CP, Poulsen I, Kammersgaard LP, Siebner HR. Alterations in the brain's connectome during recovery from severe traumatic brain injury: protocol for a longitudinal prospective study. BMJ Open. 2017 Jun 14;7(6):e016286. doi: 10.1136/bmjopen-2017-016286. PMID 28615277
- [Result] Andreasen SH, Andersen KW, Conde V, Dyrby TB, Puonti O, Kammersgaard LP, Madsen CG, Madsen KH, Poulsen I, Siebner HR. Limited Colocalization of Microbleeds and Microstructural Changes after Severe Traumatic Brain Injury. J Neurotrauma. 2020 Feb 15;37(4):581-592. doi: 10.1089/neu.2019.6608. Epub 2019 Nov 20. PMID 31588844
- [Result] Andreasen SH, Andersen KW, Conde V, Dyrby TB, Puonti O, Kammersgaard LP, Madsen CG, Madsen KH, Poulsen I, Siebner HR. Two Coarse Spatial Patterns of Altered Brain Microstructure Predict Post-traumatic Amnesia in the Subacute Stage of Severe Traumatic Brain Injury. Front Neurol. 2020 Sep 4;11:800. doi: 10.3389/fneur.2020.00800. eCollection 2020. PMID 33013616